CLINICAL TRIAL: NCT01279772
Title: A Prospective Observational Study of Newly Diagnosed Diffuse Large B Cell Primary Breast Lymphomas Treated With R-CHOP With or Without Radiotherapy
Brief Title: This Trial is a Prospective Observational Study of Newly Diagnosed Diffuse Large B Cell Primary Breast Lymphomas
Acronym: IELSG33
Status: Terminated | Type: Observational
Why Stopped: due to slow accrual (only 1 patient entered)
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Other Study IDs: IELSG33
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2012-07

CONDITIONS: Diffuse Large B-Cell Lymphoma of the Breast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, the investigators propose that the addition of rituximab will lower the risk of systemic and local relapses in patients with localized PBL. Patients will be treated with 6 cycles of RCHOP-14 or RCHOP-21. The administration of radiotherapy following chemotherapy is strongly recommended, based on the findings of the retrospective IELSG study, but will be at the discretion of the treating center.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with DLBCL of the breast.
* Patients must have CD20 positive tumors.
* Stage IE or IIE.
* Must have at least one objective measurable or evaluable disease. Baseline measurements and evaluations must be obtained within 4 weeks of registration to the study.
* Patients must have an ECOG performance status 0-2.
* Patients must have adequate organ function as evidenced by the following laboratory studies ( within 2 weeks prior to registration):

  * Creatinine Clearance > 50 ml/min
  * Total bilirubin < 2.0 mg/dl and AST < 2 x upper limit of normal. If documented hepatic involvement with lymphoma, total bilirubin can be < 3 x ULN, and AST < 5 x ULN.
  * Absolute neutrophil count > 1500/mm3 and platelet count > 100,000/mm3. If documented bone marrow involvement with lymphoma, absolute neutrophil count > 500/mm3 and platelet count > 50,000/mm3.
* Patients must be age > 18 years.
* Patients must have a normal left ventricular ejection fraction to be eligible.

Exclusion Criteria:

* historical or radiographic evidence of CNS metastasis including previously treated, resected or asymptomatic brain lesions or leptomeningeal involvement.
* pregnant or breast feeding patients. Women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception.
* active infection requiring parental antibiotics.
* known HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously untreated patients with localized DLBCL of the breast.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-10

PRIMARY OUTCOMES:
local and CNS relapse rate | 12-month

SECONDARY OUTCOMES:
progression free survival | 12-month
overall survival | 5-year
overall, complete and partial response rates following RCHOP | at the end of chemotherapy